CLINICAL TRIAL: NCT05793827
Title: Evaluating Yoga Intervention-Induced Changes in Performance and Neurophysiology in Adults With Chronic Brain Injury
Brief Title: Pilot Trial for Adults With Acquired Brain Injury
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Boettcher Webb-Waring Biomedical Research Awards (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1799
Record Dates: First submitted 2023-02-13; First posted 2023-03-31 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Acquired Brain Injury; Traumatic Brain Injury; Stroke
Keywords: Yoga; Exercise; Balance; Autonomic Nervous System; Functional Near-Infrared Spectroscopy; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The principal investigator and postdoctoral fellow are exclusively responsible for assessing outcomes and both are masked to participant group membership. The participants, interventionists, and other key persons are not masked to participant group membership, but they are not involved in any of the outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adapted Hatha Yoga (Experimental)
  Interventions: Behavioral: Adapted Hatha Yoga
- Low-Impact Exercise (Active Comparator)
  Interventions: Behavioral: Low-Impact Exercise

INTERVENTIONS:
Behavioral: Adapted Hatha Yoga — Yoga includes breath work (pranayama), gentle stretching and holding of postures (asanas), and meditation (dhyana). Modifications/adaptations are incorporated so all participants can successfully complete the yoga intervention. Yoga is delivered in a standardized progression, including: focused, slow breath with movement and breathwork throughout every session; mantras, progressively challenging yoga postures (sitting, standing, and floor); and meditation
  Arms: Adapted Hatha Yoga
Behavioral: Low-Impact Exercise — This includes low-intensity exercise, which is matched to the estimated metabolic costs of yoga, 2.5 Metabolic Equivalent of Task (MET). Sessions include warm up, cool down, and five, 10-minute exercise stations, (e.g., walking, balance, resistance bands, weight-bearing exercise, and core work). Control exercise will be prescribed between 2.0 to 3.0 METs, equating to 30 to 40% heart rate reserve. Heart rate zones are calculated for each participant and monitored to ensure proper intensity
  Arms: Low-Impact Exercise

SUMMARY:
This pilot study will compare a yoga program to a non-yoga exercise program in adults with brain injuries. The investigators will measure possible improvements in balance and heartrate. The investigators also plan to measure changes in brain function and link balance and/or heartrate improvements to changes in brain function. Ideally, this work will create a foundation for a larger-scale study.

DETAILED DESCRIPTION:
Background and Significance: Each year, an estimated 2.9 million Americans sustain brain injuries that result in emergency department visits, hospitalizations, and death. Although there are many treatment strategies in the early weeks and months after brain injury, millions of individuals live with residual disability. This residual, chronic disability often includes significant impairments and decreased brain function. Two prominent and interconnected impairments - poor balance and autonomic nervous system (ANS) dysfunction - can increase fall risk, decrease quality of life, and increase mortality. In adults with brain injury, ANS dysfunction is characterized by hyper-activation of the sympathetic nervous system, which can have damaging or even fatal impact on internal organs. To date, there are exceedingly few options for addressing these types of impairments or improving brain function in adults with chronic brain injury. However, community-based and holistic interventions, like hatha yoga, may be highly effective for simultaneously addressing balance and ANS impairments and may also improve brain function. Hatha yoga incorporates movements that improve balance, uses breathwork that may stabilize sympathetic and parasympathetic nervous system activity, can be adapted for individual needs, and has enhanced brain function in healthy adults. Despite this, there are few empirical studies investigating yoga for individuals with brain injury. To resolve this, the research team and investigator have conducted two yoga and brain injury feasibility studies and confirmed that recruitment, retainment, intervention, and neuroimaging procedures are feasible. In these studies, the investigators have found significant improvements in balance after yoga and preliminary evidence of improved brain function, even in the absence of measurable balance improvement. Finally, there is growing evidence that exercises, like yoga, can improve ANS function by regulating sympathetic and parasympathetic activity in healthy adults, suggesting significant potential for adults with chronic brain injury.

Project Objectives: Given feasibility study success and promising early findings. The investigators will conduct a pilot randomized control trial comparing 8-weeks of group yoga to 8-weeks of active control exercise in 48 adults with chronic brain injury. The investigators will test for improvements in balance and in ANS function using heart-rate variability (HRV) monitoring. The investigator will explore intervention-induced changes in brain function by evaluating intrinsic functional connectivity, using resting-state functional magnetic resonance imaging (rs-fMRI) and task-dependent neural activation, using a proxy of neural activity - oxygenated hemoglobin (HbO) - as measured with functional near-infrared spectroscopy (fNIRS) during concurrent balance tasks. Finally, if the investigators observe functional improvements in balance or ANS function and measurable changes in brain function, the investigator will then complete exploratory analyses to link functional improvements to changes in brain function.

ELIGIBILITY:
Inclusion Criteria:

* Sustained acquired brain injury at least 6 months prior
* Self-reported balance impairment of moderate or greater, via the Neurobehavioral Symptom Inventory
* Standard fMRI safety screening for MRI components only (participants can complete other study components if they are ineligible or unwilling to complete MRI)

Exclusion Criteria:

* Sustained acquired brain injury within past 6 months
* Self-reported mild balance impairment or no balance impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Standing Balance at 2 Months | Baseline is 2-3 weeks before yoga or exercise sessions begin; post-intervention is within 2 weeks of the last yoga or exercise session, or ~ 2 months..
  Acquired using a force plate during simultaneous functional near-infrared spectroscopy
Change from Baseline in Autonomic Nervous System Function at 2 Months | Baseline is 2-3 weeks before yoga or exercise sessions begin; post-intervention is within 2 weeks of the last yoga or exercise session, or ~ 2 months.
  Acquired via heart rate variability assessment using electrocardiography
Change from Baseline in Functional Connectivity of Neural Networks at 2 Months | Baseline is 2-3 weeks before yoga or exercise sessions begin; post-intervention is within 2 weeks of the last yoga or exercise session or ~ 2 months..
  Acquired via resting state functional magnetic resonance imaging
Change from Baseline in Task-Dependent Neural Activation at 2 Months | Baseline is 2-3 weeks before yoga or exercise sessions begin; post-intervention is within 2 weeks of the last yoga or exercise session or ~ 2 months..
  Acquired pre- and post-intervention via portable functional near-infrared spectroscopy during standing balance plates with force plate.

SECONDARY OUTCOMES:
Change from Baseline in Self-Reported Quality of Life at 2 Months | Baseline is 2-3 weeks before yoga or exercise sessions begin; post-intervention is within 2 weeks of the last yoga or exercise session or ~ 2 months..
  Acquired via the Traumatic Brain Injury Quality of Life Short Form Measure on NIH Toolbox app. The NIH toolbox manual does not provide a minimum or maximum score for this measure, nor does it support interpretation of the score. However, the NIH toolbox app uses the raw score from each participant and automatically converts it into a T-Score. A publication on this measure indicates (Tulsky et al. 2016) provides guidance on how to interpret T-scores, as the T-Score Mean is 50, with a Standard Deviation of 10. T-Scores above 50 indicate that individuals are having more problems in quality of life than age- and sex-matched individuals in the general population, whereas scores below 50 indicate that they are having fewer problems.
Change from Baseline in Working Memory Performance at 2 Months | Baseline is 2-3 weeks before yoga or exercise sessions begin; post-intervention is within 2 weeks of the last yoga or exercise session, or ~ 2 months. .
  Acquired via the List Sorting Working Memory Test on the NIH Toolbox app. The NIH toolbox manual does not provide a minimum or maximum score for this measure, but score interpretations are more straightforward. The NIH toolbox app uses the raw score from each participant and automatically converts it into a T-Score, along with an age-scored standard score (higher indicates better performance) and an age-adjusted national percentile (0-100%), which shows how the participant compares to age- and sex-matched peers (higher also indicates better performance).
Change from Baseline in Inhibitory Control at 2 Months | Baseline is 2-3 weeks before yoga or exercise sessions begin; post-intervention is within 2 weeks of the last yoga or exercise session, or ~ 2 months.
  Acquired via the Flanker Inhibitory Test on the NIH Toolbox app. The NIH toolbox manual does not provide a minimum or maximum score for this measure, but score interpretations are more straightforward. The NIH toolbox app uses the raw score from each participant and automatically converts it into a T-Score, along with an age-scored standard score (higher indicates better performance) and an age-adjusted national percentile (0-100%), which shows how the participant compares to age- and sex-matched peers (higher also indicates better performance).
Change from Baseline in Cognitive Flexibility at 2 Months | Baseline is 2-3 weeks before yoga or exercise sessions begin; post-intervention is within 2 weeks of the last yoga or exercise session, or ~ 2 months.
  Acquired via the Dimensional Change Card Sort Test on the NIH Toolbox app. The NIH toolbox manual does not provide a minimum or maximum score for this measure, but score interpretations are more straightforward. The NIH toolbox app uses the raw score from each participant and automatically converts it into a T-Score, along with an age-scored standard score (higher indicates better performance) and an age-adjusted national percentile (0-100%), which shows how the participant compares to age- and sex-matched peers (higher also indicates better performance).

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn Stephens, PhD, OTR, Principal Investigator — Colorado State University
Locations (1):
- Translational Medicine Institute, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
Ideally, we will upload de-identified participant data into a public repository. We are in the process of hiring and training personnel who can fulfill this role.

REFERENCES:
- [Derived] Stephens JA, Hernandez-Sarabia JA, Sharp JL, Leach HJ, Bell C, Thomas ML, Buryznska AZ, Weaver JA, Schmid AA. Adaptive yoga versus low-impact exercise for adults with chronic acquired brain injury: a pilot randomized control trial protocol. Front Hum Neurosci. 2023 Nov 23;17:1291094. doi: 10.3389/fnhum.2023.1291094. eCollection 2023. PMID 38077184